CLINICAL TRIAL: NCT02242422
Title: Serial Changes in Lower Urinary Tract Symptoms, Urine Flow and Bladder Voiding Efficiency Following Transobturator Tape Surgery for Treatment of Female Stress Urinary Incontinence
Brief Title: Serial Changes in Micturition Symptoms, Urine Flow and Bladder Voiding Efficiency Following Transobturator Tape Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Min Chul Cho, Assistant professor, DongGuk University
Other Study IDs: MCho3
Record Dates: First submitted 2014-09-14; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- transobturator tape

SUMMARY:
The aim of this study was to identify the serial changes in lower urinary tract symptoms (LUTS), urine flow and bladder voiding efficiency after transobturator tape (TOT) surgery for treatment of female stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* women who underwent transobturator tape surgery for treatment of female stress urinary incontinence

Exclusion Criteria:

* any urinary tract infection
* pregnancy
* bladder malignancy
* postoperative follow-up of less than 12 months

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women who underwent transobturator tape surgery for treatment of female stress urinary incontinence
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Change in total overactive bladder symptom score (OABSS) after surgery | 1-week, and 1-, 3-, 6- and 12-months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Min Chul Cho, M.D., Ph.D., Principal Investigator — DongGuk University
Locations (1):
- Dongguk University ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea